CLINICAL TRIAL: NCT06459414
Title: Oropharyngeal Administration Of Colostrum For Preventing Necrotizing Enterocolitis and Late-onset Sepsis In Preterm Preterms
Brief Title: Oropharyngeal Administration Of Colostrum For Preventing Necrotizing Enterocolitis in Preterrms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Atef Abdelsattar Ibrahim, Lectuere of Pediatrics and Pediatric Clinical Nutrition, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MS-615-2022
Record Dates: First submitted 2024-04-29; First posted 2024-06-14 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interventional group recieveing Oropharyngeal Of Colostrum for 3 days (Experimental): The first interventional group will receive colostrum of their mother's breast milk through oropharyngeal route for 3 days on 1 ml/kg/day
  Interventions: Other: : Oropharyngeal Administration Of Colostrum
- Interventional group recieveing Oropharyngeal Of Colostrum for 10 days (Experimental): The second interventional group will receive colostrum of their mother's breast milk through oropharyngeal route for 10 days on 1 ml/kg/day
  Interventions: Other: : Oropharyngeal Administration Of Colostrum
- Control group recieving only the standard care (No Intervention): The control group will receive only the standard care

INTERVENTIONS:
Other: : Oropharyngeal Administration Of Colostrum — Preterm less than 34 weeks gestation will receive Oropharyngeal Colostrum for 3 days ( the first group) and for 10 days( the second group)
  Other Names: Oropharyngeal Administartion of Colostrum
  Arms: Interventional group recieveing Oropharyngeal Of Colostrum for 10 days; Interventional group recieveing Oropharyngeal Of Colostrum for 3 days

SUMMARY:
Mother's milk samples will be collected during the routine expression of milk, using a hospital-grade electric breast pump, and will be stored in the NICU breastmilk refrigerator. The research doctor will prepare the syringes for the first 24 hours of the Initial Treatment Period. For neonates in the placebo group, the milk is immediately frozen, in a separate NICU breastmilk freezer to maintain blinding, for later use when enteral feedings are started. Using sterile gloves, oral syringes will be each filled with 1 mL/kg of colostrum or normal saline 0.9% (based on group assignment), capped, and covered with a white tape as a blinding procedure. Each syringe will be labeled with the patient's name, medical record number, and the date and time of preparation. Syringes will be prepared in the same sterile manner, by the research doctor, every 24 hours.

DETAILED DESCRIPTION:
Oropharyngeal administration procedure using a standardized protocol, the doctor will provide the dosing as follows: two syringes will be warmed to room temperature. The first syringe's cap is removed and the tip of the syringe is gently placed into the neonate's mouth, alongside the right buccal mucosal tissue. The syringe tip is directed posteriorly towards the oropharynx, and the total volume (0.5 mL/kg) is slowly administered, over 20 seconds. The second syringe will be placed in the neonate's mouth in the same manner, but alongside the left buccal mucosal tissue. The entire volume (0.5 mL/kg) is administered slowly, over 20 seconds. A petite swab is used to carefully swab the right buccal mucosal tissue, followed by the left buccal mucosal tissue (≤5 seconds each side). A total volume of 1 mL/kg is administered per treatment, with buccal swabbing taking place over 10 seconds. Vital signs are carefully monitored throughout the procedure. Dosing is provided every 3 hours during the period of study.

Sample size will be 34 in each group, .

* Group A: receiving oropharyngeal colostrum for 10 days.
* Group B: control group receiving placebo for 10 days.
* Group C: receiving oropharyngeal colostrum for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with gestational age (GA) ≤ 34 weeks at birth
* Neonates who will be in admitted in the neonatal intensive care unit (NICU) within 48 hours after birth.

Exclusion Criteria:

* Any contraindication for breastfeeding as mother-related (e.g. Mothers prohibited from breastfeeding because of conditions including active tuberculosis or AIDS, treatment with radioisotopes (e.g., Iodine-131, Cobalt-60, Cesium-137) and substance abuse)
* Also any contraindication for breastfeeding as infant-related (Birth complicated with severe gastrointestinal malformations).

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-08-17 (Actual)

PRIMARY OUTCOMES:
The difference in hospital length of stay between preterm neonates who received colostrum for 3 days and those who did not receive it | 2 month
  Determination of possible protective effects of colostrum via assessing the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Iman Eiada, Principal Investigator — Professor of Pediatrics
Locations (1):
- Hoda Atef Abdelsattar Ibrahim, Cairo, Egypt